CLINICAL TRIAL: NCT04343222
Title: Control of Pain in Intravitreal Injections (COPIVIN Study): A Study Evaluating the Use of Combination Topical Anesthetic and Non-Steroidal Anti-Inflammatory Drugs (NSAIDs)
Brief Title: Control of Pain in Intravitreal Injections Using Topical NSAIDs
Acronym: COPIVIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019-0095; A536000 (Other: UW Madison); SMPH/OPHTHAL&VIS SCI/GEN (Other: UW Madison)
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2020-09

CONDITIONS: Intravitreal Injections; IVI
Keywords: pain
MeSH Terms: conditions — Pain | interventions — bromfenac; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A: Bromfenac then Artificial Tears (Experimental): Participant receives 1 drop of topical Bromfenac 0.09% 30 minutes prior to the injection and then 1 drop of an artificial tear eye drop immediately after the injection and wash.
  Interventions: Drug: Bromfenac; Drug: Artificial tears
- Group B: Artificial Tears then Bromfenac (Experimental): Participant receives 1 drop of an artificial tear eye drop 30 minutes prior to the injection and then 1 drop of topical Bromfenac 0.09% immediately after the injection and wash.
  Interventions: Drug: Bromfenac; Drug: Artificial tears
- Group C: Artificial Tears then Artificial Tears (Placebo Comparator): Participants receives 1 drop of an artificial tear eye drop 30 minutes prior to the injection and then 1 drop of an artificial tear eye drop immediately after the injection and wash.
  Interventions: Drug: Artificial tears

INTERVENTIONS:
Drug: Bromfenac — An NSAID used to treat eye pain and swelling
  Arms: Group A: Bromfenac then Artificial Tears; Group B: Artificial Tears then Bromfenac
Drug: Artificial tears — eye drops to lubricate the eye and maintain moisture

SUMMARY:
Intravitreal injections (IVI) are a common form of treatment for multiple retinal pathologies. The investigators hypothesize that an intervention with a topical NSAID will alleviate pain experienced at intravitreal injection (IVI) and post-IVI. 46 participants will be recruited, randomized into 1 of 3 treatment arms, and can expect to be on study for a day.

DETAILED DESCRIPTION:
Intravitreal injections are a very common form of treatment for a variety of ocular pathologies. The use of these injections has only increased given the large utility they provide. They both improved visual outcomes and provided patients an overall better quality of life. However, a problem experienced by patients who undergo these injections is the need for multiple reoccurring injections to maintain control of their disease. It has long been an issue to provide patients optimal pain relief both during and after their intravitreal injections. Topical anesthesia is often utilized through frequent rounds of proparacaine eye drops. Other providers often use Lidocaine gel or Lidocaine-soaked cotton swaps with variable results in terms of pain control. Subconjunctival lidocaine has also been utilized with variable control of pain, however patients did report anxiety with the thought of being given an additional injection.

Patient pain is subjective and difficult to objectively quantify when comparing different methods of post-injection control. One commonly employed pain rating system is the Wong-Baker FACES pain scale which has been quite successful in objectively quantifying patient discomfort. It should be noted that this scale is only reliable in a patient whom is able to understand how the scale works.

Other research studies have shown adequate to improved pain control through the use of topical non-steroidal anti-inflammatory drug (NSAID) eye drops. One study looked at the use of topical Nepafenac 0.10% on post injection pain. This study used the McGill pain assessment questionnaire, which not only quantified pain but the additional benefit of describing the nature of the pain the patient experienced.

A clinical research study looked at pain immediately and 6 hours after injection. The researchers found that when compared to the control group (artificial tears) the group who received NSAID eye drops had better pain control. In a similar study, Bromfenac, another topical NSAID eye drop, provided good pain relief post injection, setting a precedent for the use of topical NSAIDs in controlling IVI pain.

However, studies have only reported pain relief immediately and 6 hours after injection. There have not been any studies showing pain control 24 hours post injection. Furthermore, no studies to date have compared the timing of application of a topical NSAID, in the alleviation of long-term pain patients experience. Bromfenac 0.09% is the agent of choice given its previously demonstrated effectiveness in pain control and also strength when compared to other ophthalmic NSAIDs. This was demonstrated in a paper by Sheppard that compared Bromfenac with other topical NSAID eye drops and proved that it offered approximately 3-4 times higher levels of COX-2 inhibition. It has been approved by the FDA as a one time daily eye drop to reduce inflammation. It is commonly utilized following cataract surgery to help reduce intraocular inflammation. This study looks at this medication's utility to control pain following IVI, another invasive procedure. Pain control would be assessed immediately following injection, 6 hours post injection and 24 hours post injection. This will allow evaluation of Bromfenac 0.09%'s effectiveness on overall immediate pain control as well as on ocular discomfort/soreness that can often follow IVI. Additionally, two intervention groups to compare Bromfenac 0.09% instillation 30 minutes prior to IVI and instillation immediately following IVI.

The primary goal of this study is to determine if topically administered Bromfenac 0.09% eye drops can reduce the discomfort that patient experience both during and after intravitreal injections. Additionally, the effect of both pre and post injection application of topical Bromfenac 0.09% on subjective pain scores will be investigated.

This study will be a pilot study consisting of 46 participants. These participants will be selected from those that have a diagnosis requiring intravitreal injection of an anti-VEGF agent (Vascular Endothelial Growth Factor (VEGF)). Participants that have already undergone intravitreal injection at least once before will be eligible. This will serve to minimize bias from initial injection anxiety and will give participants a comparative data point (prior injection discomfort). Participants will be randomized into one of three groups, which will be known as group A, B or C. The groups will have drop regimens as follows:

* Group A: Will receive 1 drop of topical Bromfenac 0.09% 30 minutes prior to the injection and then 1 drop of an artificial tear eye drop immediately after the injection and wash.
* Group B: Will receive 1 drop of an artificial tear eye drop 30 minutes prior to the injection and then 1 drop of topical Bromfenac 0.09% immediately after the injection and wash.
* Group C: Will receive 1 drop of an artificial tear eye drop 30 minutes prior to the injection and then 1 drop of an artificial tear eye drop immediately after the injection and wash.

All labels will be removed from the bottles and the participants will be blinded to which group they belong to. The treating physicians will also be blinded to which group the participants belong to.

Immediately following the injection, each participant will be asked to rate their pain using the Wong-Baker FACES pain scale as well as the McGill Pain Questionnaire (SF-MPQ). Participants will then be given instructions and will be told to expect a call at 6 and 24 hours regarding further follow up phone questionnaires. Participants will also be provided with a phone number to contact should they have any complications (ie. discomfort, increased pain, vision changes, or any other questions). Participants will be provided with a copy of the Wong-Baker FACES pain scale and the McGill Pain Questionnaire to take home with them. Participants will be called 6 hours post-injection for further assessment of their pain using both the Wong-Baker FACES pain scale and the McGill Pain Questionnaire (SF-MPQ). At 24 hours, participants will again be contacted and their pain will be assessed one final time using both the Wong-Baker FACES pain scale and the McGill Pain Questionnaire (SF-MPQ). This will serve as the last point of data gathered from participants.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with retinal pathology requiring anti-VEGF therapy
* Previously had an IVI

Exclusion Criteria:

* History of previous eye surgery other than cataract extraction
* Herpetic eye disease
* Uncontrolled glaucoma
* Uveitis
* Acute conjunctivitis
* Pregnancy
* Known previous adverse response or contraindication to intravitreal injection, Bromfenac, or other NSAIDs.
* Keratitis including povidone-induced keratitis
* Bullous keratopathy
* Diagnosis of dry eye syndrome
* Uncontrolled diabetes
* NSAID use 3 days prior to IVI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Mititelu, MD, MPH, Principal Investigator — University of Wisconsin, Madison; Maxwell Wingelaar, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were patients with retinal disease requiring anti-VEGF therapy under the care of retinal specialists at the University of Wisconsin Hospital and Clinics.
Period: Overall Study
Arm/Group | Group A: Bromfenac Then Artificial Tears | Group B: Artificial Tears Then Bromfenac | Group C: Artificial Tears Then Artificial Tears
Started | 16 | 15 | 15
Completed | 16 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Bromfenac Then Artificial Tears | Group B: Artificial Tears Then Bromfenac | Group C: Artificial Tears Then Artificial Tears | Total
Number analyzed (Participants) | 16 | 15 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.69 (7.69) | 78.67 (9.72) | 73.40 (8.95) | 76.61 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 13 | 31
  Male | 3 | 10 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 15 | 15 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 16 | 15 | 15 | 46
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 15 | 46
Mean Number of Prior Injections [Mean (Standard Deviation); unit: injections] | 20.81 (17.40) | 17.53 (14.40) | 10.80 (12.81) | 16.48 (15.62)
Indication for Intravitreal Injection [Count of Participants; unit: Participants]
  Age-related macular degeneration | 14 | 12 | 9 | 35
  Branch Retinal Vein Occlusion | 2 | 2 | 2 | 6
  Diabetic Macular Edema | 0 | 0 | 3 | 3
  Central retinal vein occlusion | 0 | 1 | 0 | 1
  myopic degeneration | 0 | 0 | 1 | 1
anti-VEGF agent used as SOC [Count of Participants; unit: Participants] — Anti-Vascular Endothelial Growth Factor (anti-VEGF), Standard of Care (SOC)
  Participants
    bevacizumab | 8 | 8 | 9 | 25
    aflibercept | 8 | 7 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: McGill Pain Questionnaire (SF-MPQ) Scores at Baseline
Description: Assessment of topical 0.09% Bromfenac's analgesic effect pre- and post-injection in participants undergoing intravitreal injections (IVI) of anti-VEGFs as measured by the SF-MPQ. The SF-MPQ questionnaire contains 15 sensory and affective descriptors each rated on a 0-3 scale where 0 is none, 1 is mild, 2 is moderate, and 3 is severe. The total possible range of scores is 0-45 where the higher the score, the more intense the pain.
Time Frame: Baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group A: Bromfenac Then Artificial Tears | Group B: Artificial Tears Then Bromfenac | Group C: Artificial Tears Then Artificial Tears
Number analyzed (Participants) | 16 | 15 | 15
score on a scale | 0.62 [0 to 3] | 0.93 [0 to 4] | 0.53 [0 to 2]

2. Primary Outcome: McGill Pain Questionnaire (SF-MPQ) Scores at 6 Hours Post Injection
Description: as for outcome 1
Time Frame: 6 hours post injection
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group A: Bromfenac Then Artificial Tears | Group B: Artificial Tears Then Bromfenac | Group C: Artificial Tears Then Artificial Tears
Number analyzed (Participants) | 16 | 15 | 15
score on a scale | 0.50 [0 to 2] | 0.13 [0 to 1] | 0.13 [0 to 2]

3. Primary Outcome: McGill Pain Questionnaire (SF-MPQ) Scores at 24 Hours Post Injection
Description: as for outcome 1
Time Frame: 24 hours post injection
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group A: Bromfenac Then Artificial Tears | Group B: Artificial Tears Then Bromfenac | Group C: Artificial Tears Then Artificial Tears
Number analyzed (Participants) | 16 | 15 | 15
score on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

4. Primary Outcome: Wong-Baker FACES Pain Scale Scores at Baseline
Description: Assessment of topical 0.09% Bromfenac's analgesic effect pre- and post-injection in patients undergoing intravitreal injections of anti-VEGFs as measured by the Wong-Baker FACES pain scale. This scale is compromised of drawings of faces that appear to be experiencing increasing pain, from which the participant chooses their current level of pain. Scoring is defined on the scale as, "Face 0 doesn't hurt at all. Face 2 hurts just a little bit. Face 4 hurts a little bit more. Face 6 hurts even more. Face 8 hurts a whole lot. Face 10 hurts as much as you can imagine, although you don't have to be crying to have this worst pain."
Time Frame: Baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group A: Bromfenac Then Artificial Tears | Group B: Artificial Tears Then Bromfenac | Group C: Artificial Tears Then Artificial Tears
Number analyzed (Participants) | 16 | 15 | 15
score on a scale | 0.75 [0 to 2] | 1.13 [0 to 2] | 0.53 [0 to 2]

5. Primary Outcome: Wong-Baker FACES Pain Scale Scores at 6 Hours Post Injection
Description: as for outcome 4
Time Frame: 6 hours post injection
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group A: Bromfenac Then Artificial Tears | Group B: Artificial Tears Then Bromfenac | Group C: Artificial Tears Then Artificial Tears
Number analyzed (Participants) | 16 | 15 | 15
score on a scale | 0.53 [0 to 2] | 0.07 [0 to 1] | 0.13 [0 to 2]

6. Primary Outcome: Wong-Baker FACES Pain Scale Scores at 24 Hours Post Injection
Description: as for outcome 4
Time Frame: 24 hours post injection
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group A: Bromfenac Then Artificial Tears | Group B: Artificial Tears Then Bromfenac | Group C: Artificial Tears Then Artificial Tears
Number analyzed (Participants) | 16 | 15 | 15
score on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Participants will have the opportunity to report adverse events at the time of the procedure and at 6 hours and 24 hours post injection.
Arm/Group | Group A: Bromfenac Then Artificial Tears | Group B: Artificial Tears Then Bromfenac | Group C: Artificial Tears Then Artificial Tears
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
The sample size was originally powered for a difference of 1.0 on the FACES scale. Due to the clustering of results and low pain scores reported in all arms, the 95% confidence interval included zero and prevented statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT04343222/Prot_SAP_000.pdf